CLINICAL TRIAL: NCT04806789
Title: Plasma Sodium: a Predictor of Perforation in Acute Appendicitis. (The NAP-study)
Status: Completed | Type: Observational
Sponsor: Urban Fläring (Other)
Collaborators: Odense University Hospital (Other); Charite University, Berlin, Germany (Other); Red Cross War Memorial Childrens Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Urban Fläring, Associate Professor. Senior Consultant., Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: K 2021-2319
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Appendicitis; Children, Only
Keywords: Acute appendicitis; Children; Plasma Sodium
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with suspected acute appendicitis: Cohort: Children with suspected acute appendicitis. Clinical examination (including history of nausea, vomiting, temperature, information of rebound tenderness, right iliac fossa pain, duration of symptoms, gender and weight) and blood samples will be obtained at the emergency department (blood gas, C-reactive protein, neutrophiles and white blood cell count). Radiology (ultrasound and/or computed tomography) will be performed thereafter.
  Outcome measures
  Primary outcome measure: Plasma sodium. To investigate if plasma sodium is an independent predictor of perforation in children with acute appendicitis. In advance, five variables (Plasma sodium, C-reactive protein, symptom duration, age and temperature) will be included in the final multivariable analysis

SUMMARY:
This clinical prospective diagnostic accuracy study assesses plasma sodium concentration using blood gas analysis at the emergency department in children, age 1-15 years, with suspected acute appendicitis. The overall assumption is that using plasma sodium as a biomarker, a cut-off value of <136 mmol/L will differentiate perforated from non-perforated acute appendicitis. In addition, traditionally used clinical diagnostic variables as well as radiology used in the diagnosis of acute appendicitis will also be obtained. Histopathology will be used to define if the appendix is perforated or not.

DETAILED DESCRIPTION:
Background: The historical dogma that acute appendicitis always progresses to gangrene and perforation has been rejected. In addition, there is evolving evidence that medical treatment of non-perforated acute appendicitis is safe. On the other hand, perforated acute appendicitis requires appendectomy [Andersson]. Therefore, it is important to differentiate perforation from non-perforation in order to enable proper treatment.

In a pilot-study in children with acute appendicitis (n=80), plasma sodium was shown to be an independent predictor differentiating between perforated and non-perforated acute appendicitis [Lindestam]. Using plasma sodium at a cut-off value of <136 mmol/L, the odds ratio of having a perforated acute appendicitis was 31.9 (95% CI, 6.3- 161.9) with an area under the receiver operating curve of 0.93. Sensitivity and specificity were 0.87 (95 % CI 0.60-0.98) and 0.83 (95 % CI 0.72-0.91). Similar results have later been shown by another research group [Pogorelic]. Possible mechanism for lower plasma sodium among patients with perforation is higher concentration of arginin-vasopressin, which has previously been shown [Lindestam].

Methods: Participants (n=450 in total) whereof 150 in Sweden, 150 in Republic of South Africa, 50 in Germany, 50 in Denmark and 50 in Norway will be included in the study. The patients/parents will be asked for participation in the study and included after decision of surgery has been made by the attendant surgeon. At this timepoint, (i) variables from clinical examination/history (presence of right iliac fossa pain, rebound tenderness, duration of symptoms, vomiting, temperature, gender, age, weight, (ii) blood sampling: blood gas (including plasma sodium), C-reactive protein, neutrophiles, White blood cell count (obtained at the emergency department) and (iii) radiology has been obtained. No intervention is planned. These variables will also be used to calculate the Appendicitis Inflammatory Responce (AIR) score [Scott]. Thereafter, plasma sodium concentration will be added and the score will be recalculated.

After surgery, histopathology will be used to determine if the appendix is perforated or not.

ELIGIBILITY:
Inclusion Criteria:

* Children with suspected acute appendicitis

Exclusion Criteria:

* Chronic metabolic disease
* Endocrinological disease

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with suspected acute appendicitis
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Plasma sodium concentration as a predictor for perforated acute appendicitis. | Possible predictive variables will only be obtained at one occation on the day of admission to the emergency department.
  Plasma sodium will be dichotomized at 136 mmol/L. Lower concentration are hypothesized to indicate perforated acute appendicitis.

SECONDARY OUTCOMES:
Plasma sodium concentration adding precision to the diagnostic performance of "the Appendicitis Inflammatory Response (AIR) score". | Diagnostic values of interest are only obtained at one occasion on admission to the emergency department
  This score uses anthropometric and laboratory values that will be obtained on admission to the emergency department. Adding plasma sodium to these values in regression analysis to increase possibility to predict perforated acute appendicitis.

CONTACTS AND LOCATIONS:
Overall Officials: Urban Fläring, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Pediatric Perioperative Medicine and Intensive Care, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
It is likely that we will share data on request when the study is published,

REFERENCES:
- [Background] Andersson RE, Petzold MG. Nonsurgical treatment of appendiceal abscess or phlegmon: a systematic review and meta-analysis. Ann Surg. 2007 Nov;246(5):741-8. doi: 10.1097/SLA.0b013e31811f3f9f. PMID 17968164
- [Background] Lindestam U, Almstrom M, Jacks J, Malmquist P, Lonnqvist PA, Jensen BL, Carlstrom M, Krmar RT, Svensson JF, Norberg A, Flaring U. Low Plasma Sodium Concentration Predicts Perforated Acute Appendicitis in Children: A Prospective Diagnostic Accuracy Study. Eur J Pediatr Surg. 2020 Aug;30(4):350-356. doi: 10.1055/s-0039-1687870. Epub 2019 Apr 25. PMID 31022754
- [Background] Pogorelic Z, Luksic B, Nincevic S, Luksic B, Polasek O. Hyponatremia as a predictor of perforated acute appendicitis in pediatric population: A prospective study. J Pediatr Surg. 2021 Oct;56(10):1816-1821. doi: 10.1016/j.jpedsurg.2020.09.066. Epub 2020 Oct 8. PMID 33153722
- [Background] Scott AJ, Mason SE, Arunakirinathan M, Reissis Y, Kinross JM, Smith JJ. Risk stratification by the Appendicitis Inflammatory Response score to guide decision-making in patients with suspected appendicitis. Br J Surg. 2015 Apr;102(5):563-72. doi: 10.1002/bjs.9773. Epub 2015 Mar 2. PMID 25727811
- See also: Andersson — https://pubmed-ncbi-nlm-nih-gov.proxy.kib.ki.se/17180556/
- See also: Lindestam — https://pubmed-ncbi-nlm-nih-gov.proxy.kib.ki.se/31022754/
- See also: Pogorelic — https://pubmed-ncbi-nlm-nih-gov.proxy.kib.ki.se/33153722/
- See also: Scott — https://pubmed-ncbi-nlm-nih-gov.proxy.kib.ki.se/25727811/